CLINICAL TRIAL: NCT04213755
Title: Rotational Thromboelastometry During Cesarean Section as a Predictive Evaluation for Progression of Intraoperative Massive Hemorrhage in Parturients With a Potential Risk of Perioperative Hemorrhage: a Prospective Observational Study
Brief Title: ROTEM in Patients With Placenta Previa
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: ROTEM in placenta previa
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Placenta Previa; Placenta Accreta; Placenta Increta; Placenta Percreta
MeSH Terms: conditions — Placenta Previa; Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with risks of intraoperative massive bleeding: patients with risks of intraoperative massive bleeding
  Interventions: Diagnostic Test: ROTEM

INTERVENTIONS:
Diagnostic Test: ROTEM — ROTEM including INTEM, EXTEM, APTEM, and FIBTEM

SUMMARY:
The rotational thromboelastogram (ROTEM) test can be performed on patients with placenta previa/accreta/increta/percreta who have a high likelihood of massive bleeding, and the predictors can be identified by comparing the patients who actually show massive bleeding with those who do not.

Applying these predictive factors to pregnant women undergoing cesarean section after diagnosis of placenta previa/accreta/increta/percreta, it will be advantageous for the perioperative management because it is possible to select pregnant women with a factor of massive bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section under spinal anesthesia
* Placenta previa
* Placenta accreta
* Placenta increta
* Placenta percreta

Exclusion Criteria:

* Coagulopathy
* Medication with antiplatelets or anticoagulants

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women over 20 years old who are scheduled for cesarean section under spinal anesthesia after diagnosis of placenta previa/increta/percreta/accreta
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Blood loss | 1 min after finishing an operation
  Volume of intraoperative blood loss
Change of INTEM | 10 min after spinal anesthesia, 5 min after baby delivery, 1 min after finishing operation
  intrinsic pathway component
Change of EXTEM | 10 min after spinal anesthesia, 5 min after baby delivery, 1 min after finishing operation
  extrinsic pathway component
Change of APTEM | 10 min after spinal anesthesia, 5 min after baby delivery, 1 min after finishing operation
  fibrinolytic component
Change of FIBTEM | 10 min after spinal anesthesia, 5 min after baby delivery, 1 min after finishing operation
  the level of fibrinogen

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No